CLINICAL TRIAL: NCT03670745
Title: Patient-centered Approaches to Provider and Adolescent Reproductive Health Communication and Shared Decision-making
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID pandemic and issues with the APT platform hindered recruitment and participant completion of intervention surveys.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000023279
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Reproductive Behavior
MeSH Terms: conditions — Reproductive Behavior | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This project will utilize a sequential explanatory research design, with an embedded randomized controlled trial (RCT) intervention .
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-visit Planning Tool (Experimental): To determine the effectiveness an electronic self-administered pre-visit planning tool allowing adolescents to list areas of concern to support shared decision-making during an office visit. Interviews will also explore approaches to implement and evaluate such a tool.
  Interventions: Behavioral: An electronic self-administered pre-visit planning tool.
- control group (Active Comparator): Will not be receiving an electronic self-administered pre-visit planning tool.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: An electronic self-administered pre-visit planning tool. — An electronic self-administered pre-visit planning tool allowing adolescents to list areas of concern to support shared decision-making during an office visit.
  Arms: Pre-visit Planning Tool
Behavioral: Control group — No planning tool
  Arms: control group

SUMMARY:
Determine the effectiveness of an electronic self-administered pre-visit planning tool allowing adolescents to list areas of concern to support shared decision-making and communication during an office visit through a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Aim 1: Through qualitative data collection, characterize perspectives of adolescent girls and providers regarding the feasibility and acceptability of an electronic self-administered pre-visit planning tool allowing adolescents to list areas of concern to support shared decision-making and communication during an office visit. Interviews will also explore approaches to implement and evaluate such a tool.

Aim 2: Determine the effectiveness of the tool through a randomized controlled trial (RCT).

Aim 3: Synthesize outcomes, identify opportunities for improvement and plan next steps in both research, and if the tool works well, implementation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for adolescent girls: between the ages of 14-18 years old, English-speaking, and a patient of a provider affiliated with the Yale New Haven Hospital.
* Inclusion criteria for healthcare providers are: a provider the Yale New Haven Hospital who regularly sees adolescent patients.

Exclusion Criteria:

* Exclusion criteria for adolescent girls: currently pregnant, or who have an impairment that would prevent them from completing the tool and survey.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Adolescent girls between the ages of 14-18 years
Enrollment: 10 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Sexual and Reproductive Health Knowledge Scale | up to 2 weeks after appointment
  An increase in score in the self-administered survey scale measuring knowledge adapted from the World Health Organization's Illustrative Questionnaire for Surveys with Young People from baseline to testing 2 weeks after appointment.
Contraceptive intentions | up to 2 weeks after appointment
  An increase in score in the self-administered survey questions concerning intentions to use contraceptives from baseline test to test 2 weeks after appointment. Questions adapted from the World Health Organization's Illustrative Questionnaire for Surveys with Young People
Communication with provider | up to 2 weeks after appointment
  An increased score in the self-administered survey scale measuring communication with health provider on topics of concern from baseline score to testing 2 weeks after initial appointment. Scale is adapted from the World Health Organization's Illustrative Questionnaire for Surveys with Young People

SECONDARY OUTCOMES:
Sources of sexual and reproductive health knowledge | up to 2 weeks after appointment
  An increase in score in the self-administered survey questions concerning sources of sexual and reproductive health knowledge from baseline to testing 2 weeks after initial appointment. Questions adapted from the World Health Organization's Illustrative Questionnaire for Surveys with Young People

OTHER OUTCOMES:
Use and perceptions of healthcare services | up to 2 weeks after appointment
  An increase in score of the self-administered survey questions concerning other services used and perceptions of those services provided at their appointment to scores tested 2 weeks after. Questions adapted from the World Health Organization's Illustrative Questionnaire for Surveys with Young People

CONTACTS AND LOCATIONS:
Overall Officials: Marie Brault, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided